CLINICAL TRIAL: NCT00433589
Title: MINDACT (Microarray In Node-Negative and 1 to 3 Positive Lymph Node Disease May Avoid Chemotherapy): A Prospective, Randomized Study Comparing the 70-Gene Signature With the Common Clinical-Pathological Criteria in Selecting Patients for Adjuvant Chemotherapy in Breast Cancer With 0 to 3 Positive Nodes
Brief Title: Genetic Testing or Clinical Assessment in Determining the Need for Chemotherapy in Women With Breast Cancer That Involves No More Than 3 Lymph Nodes
Acronym: MINDACT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: European Organisation for Research and Treatment of Cancer - EORTC (Network)
Collaborators: Agendia (Industry); Breast International Group (Other); Roche Pharma AG (Industry); Novartis (Industry); Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EORTC-10041; 2005-002625-31 (EudraCT Number); BIG-3-04; EU-20676; NOVARTIS-EORTC-10041; ROCHE-EORTC-10041; SANOFI-AVENTIS-EORTC-10041
Record Dates: First submitted 2007-02-08; First posted 2007-02-12 (Estimated); Last update posted 2022-11-17 (Actual); Status verified 2022-11

CONDITIONS: Breast Cancer
Keywords: invasive ductal breast carcinoma; invasive lobular breast carcinoma; stage IA breast cancer; stage IB breast cancer; stage II breast cancer; estrogen receptor-positive breast cancer; progesterone receptor-positive breast cancer
MeSH Terms: conditions — Breast Neoplasms; Carcinoma, Ductal, Breast; Carcinoma, Lobular | interventions — Docetaxel; Capecitabine; Tamoxifen; Letrozole

ARMS (6):
- Chemotherapy randomization: Arm I (anthracycline-based) (Active Comparator): * FEC 100
  * Canadian CEF
  * CAF
  * FAC
  * E-CMF
  Interventions: Drug: anthracycline-based
- Chemotherapy randomization: Arm II (docetaxel and capecitabine) (Experimental): * Docetaxel
  * Capecitabine
  Interventions: Drug: docetaxel and capecitabine
- Endocrine therapy randomization: Arm I (Active Comparator): 2 years of tamoxifen followed by 5 years of letrozole
  Interventions: Drug: tamoxifen; Drug: Letrozole
- Endocrine therapy randomization: Arm II (Experimental): 7 years of letrozole
  Interventions: Drug: Letrozole
- Treatment decision randomization: Arm I (Active Comparator): chemotherapy-decision-making according to clinical criteria (using Adjuvant! Online)
  Interventions: Drug: anthracycline-based; Drug: docetaxel and capecitabine
- Treatment decision randomization: Arm II (Experimental): chemotherapy-decision-making according to genomic prognosis using the 70-gene signature
  Interventions: Drug: anthracycline-based; Drug: docetaxel and capecitabine

INTERVENTIONS:
Drug: anthracycline-based
  Arms: Chemotherapy randomization: Arm I (anthracycline-based); Treatment decision randomization: Arm I; Treatment decision randomization: Arm II
Drug: docetaxel and capecitabine
  Arms: Chemotherapy randomization: Arm II (docetaxel and capecitabine); Treatment decision randomization: Arm I; Treatment decision randomization: Arm II
Drug: tamoxifen
  Arms: Endocrine therapy randomization: Arm I
Drug: Letrozole
  Arms: Endocrine therapy randomization: Arm I; Endocrine therapy randomization: Arm II

SUMMARY:
RATIONALE: Drugs used in chemotherapy work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving more than one drug (combination chemotherapy) may kill more tumor cells. Estrogen can cause the growth of breast cancer cells. Hormone therapy using tamoxifen may fight breast cancer by blocking the use of estrogen by the tumor cells. Letrozole may fight breast cancer by lowering the amount of estrogen the body makes. Giving chemotherapy and hormone therapy after surgery may kill any tumor cells that remain after surgery. It is not yet known whether genetic testing is more effective than clinical assessment in determining the need for chemotherapy in treating breast cancer.

PURPOSE: This randomized phase III trial is studying genetic testing to see how well it works compared with clinical assessment in determining the need for chemotherapy in women with breast cancer that is either node-negative or involves no more than 3 lymph nodes.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Compare a molecular profiling approach (70-gene signature) vs usual clinical assessment in assigning adequate risk categories (and the need to receive adjuvant chemotherapy or not) to breast cancer patients with 0-3 positive lymph nodes.
* Compare the efficacy and long-term toxicities of docetaxel and capecitabine vs standard anthracycline-based chemotherapy regimens in these patients.
* Determine the best endocrine treatment strategy (i.e., letrozole for 7 years vs sequential tamoxifen for 2 years followed by letrozole for 5 years) in these patients.

Secondary

* Compare both relative (hazard ratio) and absolute (percentage at 5 years) efficacy of these regimens, in terms of disease-free survival (DFS), distant metastasis-free survival (DMFS), and overall survival (OS), in these patients.
* Determine overall estimates of efficacy (DFS, DMFS, OS) for each treatment strategy according to clinical-pathological prognosis and molecular prognosis in these patients.
* Estimate the percentage of patients receiving chemotherapy per each prognostic method.
* Identify predictive gene expression profiles of clinical response/resistance to anthracycline-based and docetaxel-capecitabine chemotherapy in these patients.
* Compare novel gene expression signatures predicting clinical response in patients treated with sequential tamoxifen-letrozole vs letrozole alone.
* Compare the OS distributions in patients treated with these regimens.
* Compare the early and late toxicities of these regimens in these patients.
* Evaluate adjuvant endocrine treatment success or failure in the subgroup of postmenopausal patients with endocrine-responsive disease.
* Compare the safety profile of these two endocrine therapy regimens in these patients.

OUTLINE: This is a partially randomized, open-label, prospective, multicenter study.

Patients with both clinical high-risk (CHR) and genomic high-risk (GHR) disease are assigned to receive chemotherapy. Patients with both clinical low-risk (CLR) and genomic low-risk (GLR) disease do not receive chemotherapy. Patients with discordant risk between the 2 decision-making tools (standard clinical-pathological criteria vs 70-gene signature criteria) are randomized to receive chemotherapy or not. Patients with HER-2 positive tumors which have both methods discordant and were randomized to no chemotherapy, can receive adjuvant trastuzumab alone or with adjuvant endocrine therapy (if hormonal receptor positive), if decided by the treating physician. Patients with HER-2 positive tumors that are classified low-risk by both methods can receive adjuvant trastuzumab alone or with adjuvant endocrine therapy (if hormonal receptor positive), if decided by the treating physician and if no issues for trastuzumab reimbursement exist in the investigator's country.

* Chemotherapy: Patients are stratified according to participating center, risk group (GHR/CLR vs GLR/CHR), hormone receptor status (estrogen receptor [ER] positive and/or progesterone receptor [PR] positive vs ER and PR negative), age (< 50 years vs at least 50 years), HER2/neu status (positive vs negative vs unknown), method of axillary evaluation (sentinel only vs dissection), and type of surgery (mastectomy vs quadrantectomy/tumorectomy). In case PR is unknown, the patient will be stratified to the hormone receptor (HR) negative group if ER is negative, and to the HR positive group if ER is positive.

Three randomizations took place:

* One randomization on the discordant groups (where clinical risk did not match genomic risk) in treatment decision (R-T).
* One randomization for patients who are candidates for chemotherapy (R-C): randomization between anthracycline based chemotherapy and taxane/capecitabine chemotherapy.
* One randomization for patients who are candidates for endocrine therapy (R-E): randomization between 2 years of tamoxifen followed by 5 years of letrozole and 7 years of letrozole.

For the treatment decision randomization, patients for whom both methods are discordant will be randomized (R-T) between chemotherapy-decision-making according to clinical criteria (using Adjuvant! Online) or chemotherapy-decision-making according to genomic prognosis using the 70-gene signature.

For the chemotherapy randomization, patients are randomized to 1 of 2 treatment arms.

* Arm I (anthracycline-based): Patients may receive 1 of the following regimens*:

  * FEC 100: Patients receive fluorouracil IV, epirubicin hydrochloride IV, and cyclophosphamide IV on day 1. Treatment repeats every 3 weeks for 6 courses.
  * Canadian CEF: Patients receive oral cyclophosphamide on days 1-14 (or IV on days 1 and 8) and epirubicin hydrochloride IV and fluorouracil IV on days 1 and 8. Treatment repeats every 4 weeks for 6 courses.
  * CAF: Patients receive cyclophosphamide IV, doxorubicin hydrochloride IV, and fluorouracil IV on day 1. Treatment repeats every 4 weeks for 6 courses.
  * FAC: Patients receive cyclophosphamide IV and doxorubicin hydrochloride IV on day 1 and fluorouracil IV on days 1 and 8. Treatment repeats every 3 weeks for 6 courses.
  * E-CMF: Patients receive epirubicin hydrochloride IV on day 1. Treatment repeats every 3 weeks for 4 courses. Patients then receive cyclophosphamide IV, methotrexate IV, and fluorouracil IV on days 1 and 8. Treatment repeats every 4 weeks for 4 courses.

NOTE: *Patients who refuse randomization may be treated with another chemotherapy regimen and still be included in the study.

* Arm II (docetaxel and capecitabine): Patients receive docetaxel IV over 1 hour on day 1 and oral capecitabine twice daily on days 1-14. Treatment repeats every 3 weeks for 6 courses.

For the endocrine therapy randomization (all postmenopausal and some premenopausal** patients who have endocrine-responsive tumors***): Patients are stratified according to participating center, risk group (GHR/CHR vs GHR/CLR vs GLR/CHR vs GLR/CLR), adjuvant chemotherapy (no vs nonrandomized vs arm I vs arm II), endocrine sensitivity (both ER and PR positive vs either ER or PR positive), age (< 50 years vs at least 50 years), HER2/neu status (positive vs negative vs unknown), method of axillary evaluation (sentinel only vs dissection), and type of surgery (mastectomy vs quadrantectomy/tumorectomy). In case PR is unknown, the patient will be stratified to the HR negative group if ER is negative, and to the HR positive group if ER is positive.

Therapy begins after prior surgery in patients who did not receive chemotherapy and after chemotherapy in those who did. Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive oral tamoxifen citrate once daily for 2 years. Patients then receive oral letrozole once daily for 5 years.
* Arm II: Patients receive oral letrozole once daily for 7 years. NOTE: *The first dose of endocrine therapy should be administered within 4 weeks following the randomization (R-E) date. If treatment has not started within 300 days after definitive surgery, the patient becomes ineligible for randomized endocrine therapy.

NOTE: **Premenopausal women (< 50 years) must undergo adequate ovarian suppression (gonadotropin releasing hormone, bilateral oophorectomy, or bilateral ovarian radiation).

NOTE: ***Patients who have endocrine-responsive tumors but refuse randomization should receive standard endocrine therapy and may remain on study.

After completion of study treatment, patients are followed annually for at least 15 years.

FINAL ACCRUAL: A total of 6,694 patients have been accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed invasive breast cancer meeting the following criteria:

  * T1, T2, or operable T3 disease
  * Zero to three positive lymph nodes and no distant metastases
  * Unilateral tumor

    * Multifocal tumors are allowed provided that they have identical histology
    * Ductal carcinoma in situ or lobular carcinoma in situ allowed
* Operable disease

  * Must have undergone breast-conserving surgery or mastectomy with either a sentinel node procedure or full axillary clearance

    * Radiotherapy is mandatory in the case of breast-conserving surgery
    * Unresectable positive deep margins and will receive adjuvant radiotherapy provided that all other margins negative allowed
* Patients eligible for inclusion in the chemotherapy randomization must meet one of the following criteria:

  * High-risk of recurrence according to both the clinical-pathological criteria and the 70-gene signature
  * High risk of recurrence according to the clinical-pathological criteria and low-risk of recurrence according to the 70-gene signature and are randomized to use the clinical-pathological criteria for chemotherapy decision
  * Low-risk of recurrence according to the clinical-pathological criteria and high-risk of recurrence according to the 70-gene signature and are randomized to use the 70-gene signature for chemotherapy decision
* Patients eligible for inclusion in the endocrine therapy randomization must meet all of the following criteria:

  * Endocrine-responsive disease
  * Hormone receptor-positive disease (estrogen receptor-positive, progesterone receptor-positive, or both)

PATIENT CHARACTERISTICS:

* Female
* WHO performance status 0-1
* Neutrophil count > 1,500/mm^3
* Platelet count > 100,000/mm^3
* Creatinine clearance at least 50 mL/min OR creatinine up to 1.5 times upper limit of normal (ULN)
* ALT and AST up to 2.5 times ULN
* Alkaline phosphatase up to 2.5 times ULN
* Bilirubin up to 2.0 times ULN
* Normal echocardiogram (ECHO) compatible with chemotherapy treatment
* No serious cardiac illness or medical condition including, but not limited to, any of the following:

  * History of documented congestive heart failure
  * High-risk uncontrolled arrhythmias
  * Angina pectoris requiring antianginal medication
  * Clinically significant valvular heart disease
  * Evidence of transmural infarction on ECG
  * Poorly controlled hypertension (e.g., systolic blood pressure [BP] > 180 mm Hg or diastolic BP > 100 mm Hg)
  * Symptomatic coronary artery disease or a myocardial infarction within the past 12 months
  * Other risk factors that contraindicate the use of anthracycline-based chemotherapy
* No serious uncontrolled infection or other serious uncontrolled disease
* No other cancer within the past 5 years except for adequately treated carcinoma in situ of the cervix, nonmelanoma skin cancer, lobular or ductal carcinoma in situ of the breast, or any invasive cancer (other than breast cancer)
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective barrier contraception
* No psychological, familial, sociological, or geographical condition that would preclude study treatment
* No psychiatric disability
* No history of uncontrolled seizures or CNS disorders
* Patients eligible for inclusion in the chemotherapy randomization must meet all of the following additional criteria:

  * LVEF normal by ECHO or MUGA
  * No prior severe hypersensitivity reaction to drugs formulated with polysorbate 80
  * Must have physical integrity of the upper gastrointestinal tract
  * Able to swallow tablets
  * No malabsorption syndrome
* No prior thromboembolic disorder, deep vein thrombosis, or pulmonary emboli (for patients eligible for inclusion in the endocrine therapy randomization)

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* No prior neoadjuvant chemotherapy, neoadjuvant endocrine therapy, or radiotherapy for primary breast cancer
* No participation in another investigational drug study within the past 4 weeks
* No systemic hormone replacement therapy (with or without progestins) for more than 3 months in duration
* Patients eligible for inclusion in the chemotherapy randomization must meet all of the following additional criteria:

  * Interval between definitive surgery and start of chemotherapy 8-18 weeks
  * No prior organ allografts requiring immunosuppressive therapy
  * No concurrent sorivudine or chemically related analogues, such as brivudine
* Patients eligible for inclusion in the endocrine therapy randomization must meet all of the following additional criteria:

  * No prior high-dose systemic corticosteroids (except as antiemetic treatment), immunotherapy, or biological response modifiers (e.g., interferon)
  * No prior adjuvant antiestrogen therapy for > 1 month immediately after surgery, radiotherapy, and/or chemotherapy
  * No hormone replacement therapy within the past 4 weeks
  * No antiestrogens (e.g., tamoxifen or raloxifen) as chemoprevention or osteoporosis treatment for breast cancer within the past 18 months
* No concurrent primary prophylaxis with filgrastim (G-CSF), sargramostim (GM-CSF), or pegfilgrastim
* No other concurrent treatment during endocrine therapy, including the following:

  * Anticancer therapy (anti-estrogens, aromatase inhibitors, chemotherapy)
  * Investigational agents
  * Raloxifene or other selective estrogen-receptor modulators
  * Hormonal contraceptives (including depot injections and implants)

    * Intrauterine devices, including progesterone-coated, allowed
  * Oral or transdermal hormonal treatments, including estrogen, progesterone, androgen, or aromatase inhibitor

    * Local vaginal (topical) estrogens with minimal systemic absorption allowed for severe vaginal dryness/dyspareunia
* Concurrent bisphosphonates allowed

Ages: 18 Years to 120 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6600 (Estimated)
Dates: Start 2007-02; Primary Completion 2020-03 (Actual); Study Completion 2020-03 (Actual)

PRIMARY OUTCOMES:
Distant metastasis-free survival at 5 years | from enrollment/randomization
  o The primary endpoint for chemotherapy versus no chemotherapy (R-T) is that the 5-year distant metastasis free survival (DMFS) of 92% will be tested (a one-sided test).
Disease-free survival (DFS) | from enrollment/randomization
  o The primary endpoint for the chemotherapy randomization (R-C) is disease free survival (DFS).
DFS | from enrollment/randomization
  The primary test for the endocrine randomization (R-E) is DFS.

SECONDARY OUTCOMES:
Proportion of patients treated with chemotherapy based on clinical prognosis compared to 70-gene signature prognosis | from enrollment
  For R-T randomization
Overall survival at 5 years | from enrollment/randomization
  For R-T randomization
DFS at 5 years | from enrollment/randomization
  For R-T randomization
Safety (early and late) | from registration
  For R-C randomization
Overall survival at 5 years | from enrollment/randomization
  For R-C randomization
DMFS at 5 years | from enrollment/randomization
  For R-C randomization
Overall survival at 5 years | from enrollment/randomization
  For R-E randomization
DMFS at 5 years | from enrollment/randomization
  For R-E randomization

CONTACTS AND LOCATIONS:
Overall Officials: Emiel Rutgers, MD, PhD, Study Chair — The Netherlands Cancer Institute; Martine Piccart-Gebhart, MD, PhD, Study Chair — Jules Bordet Institute; Fatima Cardoso, MD, Study Chair — Champalimaud Cancer Center
Locations (1):
- Netherlands Cancer Institute - Antoni van Leeuwenhoek Hospital, Amsterdam, Netherlands

REFERENCES:
- [Background] Mook S, Bonnefoi H, Pruneri G, Larsimont D, Jaskiewicz J, Sabadell MD, MacGrogan G, Van't Veer LJ, Cardoso F, Rutgers EJ. Daily clinical practice of fresh tumour tissue freezing and gene expression profiling; logistics pilot study preceding the MINDACT trial. Eur J Cancer. 2009 May;45(7):1201-1208. doi: 10.1016/j.ejca.2009.01.004. Epub 2009 Feb 14. PMID 19232484
- [Background] Cardoso F, Van't Veer L, Rutgers E, Loi S, Mook S, Piccart-Gebhart MJ. Clinical application of the 70-gene profile: the MINDACT trial. J Clin Oncol. 2008 Feb 10;26(5):729-35. doi: 10.1200/JCO.2007.14.3222. PMID 18258980
- [Background] Cardoso F, Piccart-Gebhart M, Van't Veer L, Rutgers E; TRANSBIG Consortium. The MINDACT trial: the first prospective clinical validation of a genomic tool. Mol Oncol. 2007 Dec;1(3):246-51. doi: 10.1016/j.molonc.2007.10.004. Epub 2007 Oct 22. PMID 19383299
- [Background] Mook S, Van't Veer LJ, Rutgers EJ, Piccart-Gebhart MJ, Cardoso F. Individualization of therapy using Mammaprint: from development to the MINDACT Trial. Cancer Genomics Proteomics. 2007 May-Jun;4(3):147-55. PMID 17878518
- [Background] Bogaerts J, Cardoso F, Buyse M, Braga S, Loi S, Harrison JA, Bines J, Mook S, Decker N, Ravdin P, Therasse P, Rutgers E, van 't Veer LJ, Piccart M; TRANSBIG consortium. Gene signature evaluation as a prognostic tool: challenges in the design of the MINDACT trial. Nat Clin Pract Oncol. 2006 Oct;3(10):540-51. doi: 10.1038/ncponc0591. PMID 17019432
- [Result] Viale G, Slaets L, Bogaerts J, Rutgers E, Van't Veer L, Piccart-Gebhart MJ, de Snoo FA, Stork-Sloots L, Russo L, Dell'Orto P, van den Akker J, Glas A, Cardoso F; TRANSBIG Consortium & the MINDACT Investigators. High concordance of protein (by IHC), gene (by FISH; HER2 only), and microarray readout (by TargetPrint) of ER, PgR, and HER2: results from the EORTC 10041/BIG 03-04 MINDACT trial. Ann Oncol. 2014 Apr;25(4):816-823. doi: 10.1093/annonc/mdu026. PMID 24667714
- [Result] Rutgers E, Piccart-Gebhart MJ, Bogaerts J, Delaloge S, Veer LV, Rubio IT, Viale G, Thompson AM, Passalacqua R, Nitz U, Vindevoghel A, Pierga JY, Ravdin PM, Werutsky G, Cardoso F. The EORTC 10041/BIG 03-04 MINDACT trial is feasible: results of the pilot phase. Eur J Cancer. 2011 Dec;47(18):2742-9. doi: 10.1016/j.ejca.2011.09.016. Epub 2011 Nov 1. PMID 22051734
- [Derived] Alaeikhanehshir S, Ajayi T, Duijnhoven FH, Poncet C, Olaniran RO, Lips EH, van 't Veer LJ, Delaloge S, Rubio IT, Thompson AM, Cardoso F, Piccart M, Rutgers EJT. Locoregional Breast Cancer Recurrence in the European Organisation for Research and Treatment of Cancer 10041/BIG 03-04 MINDACT Trial: Analysis of Risk Factors Including the 70-Gene Signature. J Clin Oncol. 2024 Apr 1;42(10):1124-1134. doi: 10.1200/JCO.22.02690. Epub 2024 Jan 19. PMID 38241603
- [Derived] Piccart M, van 't Veer LJ, Poncet C, Lopes Cardozo JMN, Delaloge S, Pierga JY, Vuylsteke P, Brain E, Vrijaldenhoven S, Neijenhuis PA, Causeret S, Smilde TJ, Viale G, Glas AM, Delorenzi M, Sotiriou C, Rubio IT, Kummel S, Zoppoli G, Thompson AM, Matos E, Zaman K, Hilbers F, Fumagalli D, Ravdin P, Knox S, Tryfonidis K, Peric A, Meulemans B, Bogaerts J, Cardoso F, Rutgers EJT. 70-gene signature as an aid for treatment decisions in early breast cancer: updated results of the phase 3 randomised MINDACT trial with an exploratory analysis by age. Lancet Oncol. 2021 Apr;22(4):476-488. doi: 10.1016/S1470-2045(21)00007-3. Epub 2021 Mar 12. PMID 33721561
- [Derived] Delaloge S, Piccart M, Rutgers E, Litiere S, van 't Veer LJ, van den Berkmortel F, Brain E, Dudek-Peric A, Gil-Gil M, Gomez P, Hilbers FS, Khalil Z, Knox S, Kuemmel S, Kunz G, Lesur A, Pierga JY, Ravdin P, Rubio IT, Saghatchian M, Smilde TJ, Thompson AM, Viale G, Zoppoli G, Vuylsteke P, Tryfonidis K, Poncet C, Bogaerts J, Cardoso F; MINDACT investigators and the TRANSBIG Consortium. Standard Anthracycline Based Versus Docetaxel-Capecitabine in Early High Clinical and/or Genomic Risk Breast Cancer in the EORTC 10041/BIG 3-04 MINDACT Phase III Trial. J Clin Oncol. 2020 Apr 10;38(11):1186-1197. doi: 10.1200/JCO.19.01371. Epub 2020 Feb 21. PMID 32083990
- [Derived] Cardoso F, van't Veer LJ, Bogaerts J, Slaets L, Viale G, Delaloge S, Pierga JY, Brain E, Causeret S, DeLorenzi M, Glas AM, Golfinopoulos V, Goulioti T, Knox S, Matos E, Meulemans B, Neijenhuis PA, Nitz U, Passalacqua R, Ravdin P, Rubio IT, Saghatchian M, Smilde TJ, Sotiriou C, Stork L, Straehle C, Thomas G, Thompson AM, van der Hoeven JM, Vuylsteke P, Bernards R, Tryfonidis K, Rutgers E, Piccart M; MINDACT Investigators. 70-Gene Signature as an Aid to Treatment Decisions in Early-Stage Breast Cancer. N Engl J Med. 2016 Aug 25;375(8):717-29. doi: 10.1056/NEJMoa1602253. PMID 27557300
- See also: Clinical trial summary from the EORTC website — https://www.eortc.org/research_field/clinical-detail/10041/